CLINICAL TRIAL: NCT03232151
Title: C-arm Cone Beam CT Perfusion Guided Cerebrovascular Interventions Evaluating Predictability and Accuracy for the Treatment of Acute Cerebral Ischemia in the Angiography Suite
Brief Title: C-arm Cone Beam CT Perfusion Guided Cerebrovascular Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2015-0482; 1U01EB021183-01 (NIH); A539300 (Other: UW Madison); SMPH\RADIOLOGY\RADIOLOGY (Other: UW Madison); Protocol Version 3/27/2020 (Other: UW Madison)
Record Dates: First submitted 2017-07-18; First posted 2017-07-27 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: Single center, open label, single-arm, pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- C-ARM CBCT (Experimental): A C-arm CBCT evaluation with SMART RECON novel software for the rapid assessment of time-resolved CT angiogram and CT perfusion.
  Interventions: Diagnostic Test: C-Arm Cone Beam Computed Tomography

INTERVENTIONS:
Diagnostic Test: C-Arm Cone Beam Computed Tomography — C-ARM CBCT angiogram and CBCT perfusion imaging using prototype software (SMART-RECON) can rapidly and accurately assess the cerebral blood flow maps in the setting of decreased blood flow to the brain (ischemic cerebrovascular events). This rapid assessment would eliminate the need for the patient to be imaged in another scanner and be subsequently transported again to another room; all anatomic and physiologic imaging would occur in the angiography suite.
  Other Names: C-ARM CBCT

SUMMARY:
The overarching objective of our proposal is to develop a One-Stop-Shop imaging using the available C-arm Cone-Beam Computed Tomography (CBCT) data acquisition systems currently widely available worldwide in interventional angiography suites to enable acute ischemic stroke patients to be imaged, triaged, treated, and assessed using a single modality in one room.

DETAILED DESCRIPTION:
This is an evaluation to determine the efficacy of the use of C-arm CBCT with SMART RECON novel software for the rapid assessment of time-resolved CTA and CT perfusion in the setting of ischemic cerebrovascular events. As a leading center for the treatment of cerebrovascular disease in the Midwest as well as being one of the first Comprehensive Stroke Centers in the United States we have a large potential patient group to assess.

The pilot plan is to compare conventional CT/CTA/CTP acquired during the clinical work up with C-arm CBCT/CTA/CTP acquired in the angiography suite at initiation of therapy. The C-arm CBCT acquisition provides whole brain coverage (compared to only 8 cm brain coverage with conventional CT) with less radiation and higher resolution; the CT perfusion maps obtained using C-arm CBCT and new reconstruction algorithms provides better perfusion maps.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute ischemic stroke presenting within 8 hours of onset
2. Patients that present with a large artery occlusion
3. Adults 18 years of age or older.
4. Women of childbearing potential must not be pregnant.
5. National Institutes of Health Stroke Scale (NIHSS) of >5
6. No severe co-morbidities

Exclusion Criteria:

1. Women that are pregnant
2. History of severe renal disease (e.g. stage 4-5)
3. History of renal transplant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Percent of C-arm Cone Beam CT scans that detect Hyperemia or Oligemia compared to Standard of Care conventional CT | 1 study visit up to 1 hour
  To demonstrate device feasibility for phase 2 of this study, the investigators need to demonstrate that the presence of hyperemia or oligemia detected with standard of care conventional CT is also detected to a clinically acceptable degree with C-arm Cone Beam CT.

SECONDARY OUTCOMES:
Optimization of One-Stop-Shop Imaging | Up to 24 months
  Data collected will be used to optimize C-arm CBCT imaging parameters, data acquisition methods and contrast dose.
Analysis of Perfusion Parameters from One-Stop-Shop Perfusion Maps | Up to 24 months
  Local perfusion parameters on image slices will be measured and compared against the corresponding measurements from diagnostic CTP measurements.
Analysis of ROIs from One-Stop-Shop Perfusion Maps | Up to 24 months
  Standard deviations for a variety of regions of interest (ROIs) on image slices will be measured and compared against the corresponding measurements from diagnostic CTP measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Aagaard-Kienitz, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No